CLINICAL TRIAL: NCT01611376
Title: Comparison of Cardiac Output Derived From Flotrac/Vigileo and Impedance Cardiography During Major Abdominal Surgery
Brief Title: Impedance Cardiography During Major Abdominal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inje University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICG-01-Choe
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2012-05

CONDITIONS: Abdominal Surgery
Keywords: impedance cardiography; Flotrac/Vigileo; cardiac output
MeSH Terms: interventions — Cardiography, Impedance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Niccomo™ (Medis, Ilmenau, Germany) impedance cardiography

SUMMARY:
The investigators validated ICG's(impedance cardiography) usefulness during the abdominal surgery, by comparing it with FloTrac/Vigileo™ (Edwards Lifesciences,Irvine, CA, USA)

DETAILED DESCRIPTION:
Intrathoracic structures have relatively constant resistance except the influence of changing diameter of aorta. Great vessels in thorax has the lowest resistance, and their diameter changes by the beats of the heart. As their diameter increases, their resistance decreases. ICG measures the difference between the resistances caused by heartbeats, and calculates cardiac output.

But during the surgery, there are many interfering electrical currents made by electro cautery, patient positioning, and internal organ handling. Therefore, it has been thought that ICG is not a valid tool for measuring cardiac output during the surgery.

The investigators validated ICG's usefulness during the surgery, by comparing it with Floctac/Vigileo.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open gastrectomy with arterial line
* ASA 1 & 2

Exclusion Criteria:

* severe valve disease
* severe lung disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Cardiac output
  Cardiac output will be measured using an ICG and compared with cardiac output measured using Flotrac/vigileo

CONTACTS AND LOCATIONS:
Overall Officials: Won Joo Choe, Study Chair — Ilsan-Paik Hospital; Jun Hyun Kim, Study Director — Ilsan-Paik Hospital; Kyung woo Kim, Principal Investigator — Ilsan-Paik Hospital
Locations (1):
- Ilsan Paik hospital, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Result] Kim JY, Kim BR, Lee KH, Kim KW, Kim JH, Lee SI, Kim KT, Choe WJ, Park JS, Kim JW. Comparison of cardiac output derived from FloTrac/Vigileo and impedance cardiography during major abdominal surgery. J Int Med Res. 2013 Aug;41(4):1342-9. doi: 10.1177/0300060513487649. Epub 2013 Jun 26. PMID 23803309